CLINICAL TRIAL: NCT01352650
Title: Induction Therapy With Decitabine and Plerixafor Priming for Patients ≥ 60 Years With Acute Myeloid Leukemia
Brief Title: Decitabine and Plerixafor in Elderly Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1104011617
Record Dates: First submitted 2011-04-18; First posted 2011-05-12 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — plerixafor; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Cohort 1A (Active Comparator): Cycle 1: decitabine 20 mg/m2 IV daily for a 1-hour infusion on days 1-10 Cycle 2: decitabine 20 mg/m2 IV daily for a 1-hour infusion on days 1-10 + plerixafor 320 mcg/kg IV on days 1-5 Cycle 3: decitabine 20 mg/m2 IV daily for a 1-hour infusion on days 1-10 Cycle 4: decitabine 20 mg/m2 IV daily for a 1-hour infusion on days 1-10 + plerixafor 320 mcg/kg IV on days 1-5
  Interventions: Drug: plerixafor; Drug: decitabine
- Cohort 1B (Active Comparator): Cycle 1: decitabine 20 mg/m2 IV daily for a 1-hour infusion on days 1-10 + plerixafor 320 mcg/kg IV on days 1-5 Cycle 2: decitabine 20 mg/m2 IV daily for a 1-hour infusion on days 1-10 Cycle 3: decitabine 20 mg/m2 IV daily for a 1-hour infusion on days 1-10 + plerixafor 320 mcg/kg IV on days 1-5 Cycle 4: decitabine 20 mg/m2 IV daily for a 1-hour infusion on days 1-10
  Interventions: Drug: plerixafor; Drug: decitabine
- Cohort 2A (Active Comparator): Cycle 1: decitabine 20 mg/m2 IV daily for a 1-hour infusion on days 1-10 Cycle 2: decitabine 20 mg/m2 IV daily for a 1-hour infusion on days 1-10 + plerixafor 540 mcg/kg IV on days 1-5 Cycle 3: decitabine 20 mg/m2 IV daily for a 1-hour infusion on days 1-10 Cycle 4: decitabine 20 mg/m2 IV daily for a 1-hour infusion on days 1-10 + plerixafor 540 mcg/kg IV on days 1-5
  Interventions: Drug: plerixafor; Drug: decitabine
- Cohort 2B (Active Comparator): Cycle 1: decitabine 20 mg/m2 IV daily for a 1-hour infusion on days 1-10 + plerixafor 540 mcg/kg IV on days 1-5 Cycle 2 decitabine 20 mg/m2 IV daily for a 1-hour infusion on days 1-10 Cycle 3: decitabine 20 mg/m2 IV daily for a 1-hour infusion on days 1-10 + plerixafor 540 mcg/kg IV on days 1-5 Cycle 4 decitabine 20 mg/m2 IV daily for a 1-hour infusion on days 1-10
  Interventions: Drug: plerixafor; Drug: decitabine
- Cohort 3A (Active Comparator): Cycle 1: decitabine 20mg/m2 IV daily for a 1-hour infusion on days 1-10 Cycle 2: decitabine 20mg/m2 IV daily for a 1-hour infusion on days 1-10 + plerixafor 810 mcg/kg IV on days 1-5 Cycle 3: decitabine 20mg/m2 IV daily for a 1-hour infusion on days 1-10 Cycle 4: decitabine 20mg/m2 IV daily for a 1-hour infusion on days 1-10 + plerixafor 810 mcg/kg IV on days 1-5
  Interventions: Drug: plerixafor; Drug: decitabine
- Cohort 3B (Active Comparator): Cycle 1: decitabine 20mg/m2 IV daily for a 1-hour infusion on days 1-10 + plerixafor 810 mcg/kg IV on days 1-5 Cycle 2: decitabine 20mg/m2 IV daily for a 1-hour infusion on days 1-10 Cycle 3: decitabine 20mg/m2 IV daily for a 1-hour infusion on days 1-10 + plerixafor 810 mcg/kg IV on days 1-5 Cycle 4: decitabine 20mg/m2 IV daily for a 1-hour infusion on days 1-10
  Interventions: Drug: plerixafor; Drug: decitabine

INTERVENTIONS:
Drug: plerixafor — Cohort 1 will receive plerixafor at a dose of 320 mcg/kg, cohort 2 will receive plerixafor at a dose of 540 mcg/kg and cohort 3 will receive plerixafor at a dose of 810 mcg/kg. Schedule A will receive plerixafor on the 2nd and 4th cycles and Schedule B will receive plerixafor on the 1st and 3rd cycles of treatment.
  Other Names: MOZOBIL
Drug: decitabine — decitabine will be given to all cohorts/schedules at 20 mg/m2 IV daily for a 1-hour infusion on days 1-10 for all cycles
  Other Names: Dacogen

SUMMARY:
The hypothesis of this proposal is that combining plerixafor, an inhibitor of stromal cell derived factor - 1α (SDF-1α), with decitabine, a DNA methyltransferase inhibitor, as induction and postremission therapy for older patients with Acute Myeloid Leukemia (AML) will improve treatment outcomes via mobilization of leukemia stem cells and alteration of the pharmacodynamics of decitabine. The protocol will establish the safety and feasibility of combining two different doses of plerixafor with a fixed dose and schedule of decitabine.

ELIGIBILITY:
Inclusion Criteria:

* Unequivocal pathologic diagnosis of AML (≥ 20% blasts in the bone marrow based on WHO criteria) excluding: i) acute promyelocytic leukemia t(15;17)(q22;q12); PML-RARA; ii)acute myeloid leukemia with t(8;21)(q22;q22); RUNX1-RUNXT1; iii) acute myeloid leukemia with inv(16)(p13.1;q22) or t(16;16)(p13.1;q22); CBFB-MYH11.
* AML patients with an antecedent hematologic disorder or myelodysplastic syndrome (MDS)are eligible for treatment on this trial provided that they have not received prior treatment with decitabine or prior cytotoxic treatment for AML.
* AML patients with therapy-related myeloid neoplasms (t-MN) are eligible if they have not received chemotherapy (not including hormonal therapy) for their primary malignancy or disorder for >6 months.
* Age ≥ 60 years.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior treatment with decitabine
* Prior treatment with plerixafor
* Ongoing treatment for another malignancy.
* Patients with good-risk molecular or cytogenetics features
* Patient has a medical condition or illness considered by the investigator to constitute an unwarranted high risk for investigational drug treatment.
* Patient has a psychiatric disorder or altered mental status that would preclude understanding of the informed consent process and/or completion of the necessary studies.
* Patient has an inability or unwillingness, in the opinion of the investigator, to comply with the protocol requirements.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2011-06-17 (Actual); Primary Completion 2016-12-27 (Actual); Study Completion 2016-12-27 (Actual)

PRIMARY OUTCOMES:
response to treatment | after every cycle (every month) - average subject will be on study for 4-6 months
  blood and bone marrow testing will be done to determine response to treatment every month

CONTACTS AND LOCATIONS:
Overall Officials: Gail Roboz, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roboz GJ, Ritchie EK, Dault Y, Lam L, Marshall DC, Cruz NM, Hsu HC, Hassane DC, Christos PJ, Ippoliti C, Scandura JM, Guzman ML. Phase I trial of plerixafor combined with decitabine in newly diagnosed older patients with acute myeloid leukemia. Haematologica. 2018 Aug;103(8):1308-1316. doi: 10.3324/haematol.2017.183418. Epub 2018 May 3. PMID 29724902
- [Derived] Allan JN, Roboz GJ, Askin G, Ritchie E, Scandura J, Christos P, Hassane DC, Guzman ML. CD25 expression and outcomes in older patients with acute myelogenous leukemia treated with plerixafor and decitabine. Leuk Lymphoma. 2018 Apr;59(4):821-828. doi: 10.1080/10428194.2017.1352089. Epub 2017 Jul 18. PMID 28718760
- See also: Related Info — http://www.cornellmedicine.com/trials/cancer-and-blood-disorders/